CLINICAL TRIAL: NCT07165106
Title: Comparison of the Effects of Resistance and Aerobic Exercises Added to Conventional Rehabilitation Program on Walking and Sarcopenic Parameters in Patients With Sarcopenic Parkinson's Disease
Brief Title: Effects of Resistance and Aerobic Exercises on Walking and Sarcopenic Parameters in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nedime Seven Tas, Principal Investigator, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AhiEvranUERH-FTR-NST-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: PARKINSON DISEASE (Disorder); Sarcopenia
Keywords: rehabilitation; sarcopenia; exercises
MeSH Terms: conditions — Parkinson Disease; Sarcopenia; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Intervention Model Description: Three groups with a exercise control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional rehabilitation + Aerobic exercise (Experimental): Participants will receive a standard conventional rehabilitation program combined with supervised aerobic exercise training (e.g., treadmill ) according to guideline-based frequency, intensity, and duration.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Conventional Rehabilitation
- Conventional rehabilitation + Resistance exercises (Experimental): Participants will receive a standard conventional rehabilitation program combined with supervised resistance exercise training targeting major muscle groups with free weights or elastic bands.
  Interventions: Behavioral: Resistance Exercise; Behavioral: Conventional Rehabilitation
- Conventional rehabilitation (Active Comparator): Participants will receive only the standard conventional rehabilitation program without any additional aerobic or resistance exercise.
  Interventions: Behavioral: Conventional Rehabilitation

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants in this group will receive conventional rehabilitation in combination with supervised treadmill-based aerobic exercise three times per week for 6 weeks. Each exercise session will consist of a 5-minute warm-up, a 15-minute main exercise phase, and a 5-minute cool-down. Walking speed will be individualized based on participant tolerance and progressively increased under clinical supervision. Exercise intensity will be monitored using the modified Borg Rating of Perceived Exertion (scale 6-20).
  Weeks 1-2: Main exercise at Borg 10-11 (light-moderate).
  Weeks 3-4: Main exercise at Borg 11-12 (moderate).
  Weeks 5-6: Main exercise at Borg 12-13 (moderate-high).
  Cardiorespiratory responses will be monitored during all sessions, and treadmill speed will be gradually adjusted in accordance with improvements in exercise tolerance while maintaining safety.
  Other Names: Aerobic training
  Arms: Conventional rehabilitation + Aerobic exercise
Behavioral: Resistance Exercise — Participants in this arm will receive conventional rehabilitation combined with supervised resistance training using elastic bands, 3 times per week for 6 weeks. Exercises target major upper- and lower-limb and hip muscles. Each exercise is performed for 3 sets of 10 repetitions with 60-90 seconds rest. Initial band tension is set at the highest tolerable level and progressively increased. The program includes shoulder press, biceps curl, triceps extension, seated leg extension, calf raise, and lateral band walk. All sessions are supervised, emphasizing correct posture, controlled full range of motion, and avoidance of compensatory movements. Patients are guided with verbal and visual cues when necessary.
  Other Names: Resistance training
  Arms: Conventional rehabilitation + Resistance exercises
Behavioral: Conventional Rehabilitation — Participants in this group will receive conventional rehabilitation only, 5 days per week, 1 hour per day, for 6 weeks. The program includes upper and lower limb range of motion exercises, stretching, walking practice, balance and coordination training, proprioceptive exercises, posture correction, obstacle crossing, and turning in place. All sessions are delivered under clinical supervision, with emphasis on correct posture, safety, and full range of motion
  Other Names: Conventional therapy

SUMMARY:
The aim of this study was to investigate the effects of resistance and aerobic exercises on the following outcomes in patients with sarcopenic Parkinson's disease: Timed Up and Go Test (TUG), gait speed, Short Physical Performance Battery (SPPB), handgrip strength, Five-Times Sit-to-Stand Test, and MDS-UPDRS Part II scores.

DETAILED DESCRIPTION:
Female and male patients aged between 40 and 85 years, who meet the inclusion criteria, will be recruited from the Outpatient Clinic of Physical Medicine and Rehabilitation (PMR), Ahi Evran University Kırşehir Training and Research Hospital. A total of 30 participants will be enrolled in the study.

This is a prospective, randomized, controlled trial. Assessments will be performed at baseline (week 0), at the end of treatment (week 6), and at follow-up (week 12). Outcome measures will include:

Handgrip strength Timed Up and Go Test (TUG) 4-meter gait speed test Short Physical Performance Battery (SPPB) Five-Times Sit-to-Stand Test (5CST) MDS-UPDRS Part II questionnaire

In addition, at baseline, ultrasonographic measurement of anterior thigh muscle thickness will be performed. This value, expressed in millimeters, will be divided by the body mass index (BMI) to calculate the STAR (Sonographic Thigh Adjustment Ratio) index.Participants will be randomized into three treatment groups:

Group 3 (Conventional Rehabilitation Program):

Patients will receive a standard physical therapy program, 5 days per week, for 1 hour per session. The protocol will include range of motion exercises for upper and lower extremities, stretching, walking, balance and coordination training, proprioceptive exercises, postural exercises, obstacle negotiation training, and turning-in-place exercises.

Group 2 (Conventional Rehabilitation + Resistance Training):

In addition to the conventional program, patients will perform resistance exercises for major muscle groups of the upper and lower extremities using elastic resistance bands, 3 days per week.

Group 1 (Conventional Rehabilitation + Treadmill Training):

In addition to the conventional program, patients will undergo treadmill exercise consisting of a 5-minute warm-up, 15 minutes of main exercise, and 5 minutes of cool-down. Walking speed will be individually adjusted according to participant tolerance, and exercise intensity will be monitored using the Borg Rating of Perceived Exertion (RPE) scale. Treadmill speed will be progressively increased in subsequent sessions under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40-85 years with a clinical diagnosis of Parkinson's disease.
* Diagnosis of sarcopenia according to the EWGSOP2 criteria.
* Hoehn & Yahr stage 2-3.
* Ability and willingness to provide written informed consent according to the approved study consent form.

Exclusion Criteria:

* Failure to meet diagnostic criteria for sarcopenia.
* Hoehn & Yahr stage 1 or 4.
* History of malignancy.
* Epilepsy.
* History of cardiac pacemaker implantation.
* Presence of congestive heart failure.
* Orthopedic conditions affecting walking or balance.
* Respiratory disorders impairing exercise capacity.
* Uncontrolled hypertension.
* Inability to cooperate with study procedures.
* History of neuromuscular or vestibular disorders affecting gait or balance parameters.
* Lack of willingness to participate in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test (TUG Test) | BEFORE TREATMENT(WEEK 0),AT THE END OF TREATMENT (WEEK 6) AND AFTER TREATMENT (WEEK 12)
  The Timed Up and Go (TUG) test measures mobility by timing a participant rising from a chair, walking 3 m, turning, and sitting down. Lower values indicate better performance.
  Unit of Measure: seconds
4-Meter Walking Speed | BEFORE TREATMENT(WEEK 0),AT THE END OF TREATMENT (WEEK 6) AND AFTER TREATMENT (WEEK 12)
  Usual-pace walking speed over a 4-meter course, recorded as distance divided by time. Higher values indicate better performance.
  Unit of Measure: meters/second
Short Physical Performance Battery (SPPB) Score | BEFORE TREATMENT(WEEK 0),AT THE END OF TREATMENT (WEEK 6) AND AFTER TREATMENT (WEEK 12)
  Composite score including balance tests, 4-meter gait speed, and repeated chair stands; range 0 (worst) to 12 (best). Higher scores indicate better performance.
  Unit of Measure: score (0-12)
Handgrip Strength | BEFORE TREATMENT(WEEK 0),AT THE END OF TREATMENT (WEEK 6) AND AFTER TREATMENT (WEEK 12)
  Maximal isometric handgrip strength of the dominant hand measured with a handheld dynamometer. Higher values indicate better strength
Five Times Chair Stand Test | BEFORE TREATMENT(WEEK 0),AT THE END OF TREATMENT (WEEK 6) AND AFTER TREATMENT (WEEK 12)
  Time (in seconds) to rise from a chair and sit back down five consecutive times without using arms. Lower values indicate better performance.
  Unit of Measure: seconds

SECONDARY OUTCOMES:
MDS-UPDRS Part II: Motor Aspects of Experiences of Daily Living | BEFORE TREATMENT(WEEK 0),AT THE END OF TREATMENT (WEEK 6) AND AFTER TREATMENT (WEEK 12)
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II assesses the motor aspects of experiences of daily living in patients with Parkinson's disease. It is a patient-reported questionnaire evaluating difficulties in speech, saliva and drooling, chewing and swallowing, handwriting, dressing, hygiene, turning in bed, walking and balance, tremor, and fine motor tasks. Each item is scored on a 0-4 scale, with higher scores reflecting greater disability. The total score provides an index of motor impairment in daily life activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No